CLINICAL TRIAL: NCT06215339
Title: The Effect of Hemodialysis Patients' Attitudes Towards Diet Therapy on Dialysis Symptoms: A Randomized Controlled Clinical Study
Brief Title: Diet Therapy in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilan aktepe coşar (Other)
Responsible Party: Sponsor-Investigator, Dilan aktepe coşar, Lecturer, Gümüşhane Universıty
Organization: Gümüşhane Universıty (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hm20231001
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Hemolysis; Diet; Symptoms and Signs; Healthy
Keywords: Hemolysis; Diet; Healthy; Symptoms and Signs
MeSH Terms: conditions — Hemolysis; Signs and Symptoms | interventions — Population Groups; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: using G*Power 3.1.9.2. The sample size was deemed sufficient (experiment=30; control=30), and the study was concluded. Participants were selected using a lottery method, and data were collected through a singleblind randomization process.
Masking Description: While the patients were randomized; In order to keep the possibility of being affected by each other at a minimum level, the study was continued with the same application group in the same session group. For example; It's like working only with the robot cat group in the 08:00-12:00 session group on Mondays. In order to reduce the possibility of selection bias due to sample selection, "single-stage cluster type random sampling", which is a subtype of random sampling, was used. In addition, before the study, patients were informed about the study and their consent was obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group where diet education is given (Experimental): Patients in the experimental group were given face-to-face diet education by the researcher in the waiting room for approximately 15 minutes and an "Information Brochure" was given.
  Pre-training (pre-test) for hemodialysis patients Data collection tools were applied. All data collection tools were applied to these patients, except for the structured Patient Information Form for post-training measurements (intermediate measurement) 1 month after the training was given.
  Interventions: Behavioral: diet therapy training
- Control group (No Intervention): No treatment was performed on hemodialysis patients in this group. Only data collection forms were applied to the patients before the study (pretest), at the 1st week (intermediate measurement/1st measurement) and at the end of the study. (8th week) 3 times in total for 8 weeks.

INTERVENTIONS:
Behavioral: diet therapy training — diet education
  Other Names: Group without diet education
  Arms: group where diet education is given

SUMMARY:
This study determined the effect of dietary education given to hemodialysis patients on dietary treatment and symptoms.

DETAILED DESCRIPTION:
Diet therapy is a part of the treatment of hemodialysis patients. In order for the treatment to be effective, it is necessary to comply with the diet. Non-compliance with diet treatment affects the symptoms experienced by the patient, resulting in morbidity, low quality of life and mortality. Knowing patients' compliance with diet therapy is important in ensuring symptom control. The aim of this study is to determine the effect of diet therapy on symptom management in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

Being ≥18 years old,

* Agreeing to participate in the research,
* Being literate,
* Being able to communicate verbally,
* Receiving outpatient HD treatment three sessions a week at the same institution,
* No impairment in mental and cognitive functions,
* Has been receiving HD treatment for at least three months (to be defined as a chronic HD program)

Exclusion Criteria:

* Refusal to participate in the research,
* Being on peritoneal dialysis,
* Being diagnosed with a psychiatric disorder diagnosed by a psychiatrist,
* The general condition (hemodynamically) is unstable (heart rate < 100 mm/Hg or diastolic BP< 60 mm/Hg),

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Hemodialysis Patients' Attitude Scale Towards Diet Therapy (HDTO)" | 4 week
  "HDTÖ" (HD Dietary Attitude Scale):
  Each item is scored as 1-Strongly Agree, 2-Agree, 3-Disagree, 4-Strongly Disagree. The scale comprises three sub-dimensions:

SECONDARY OUTCOMES:
"Dialysis Symptom Index (DSI)" | 4 week
  this scale assesses the emotional and physical symptoms of dialysis patients and the severity of these symptoms, consisting of a total of 30 items

CONTACTS AND LOCATIONS:
Overall Officials: Dilan aktepe coşar, lecture, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gümüşhane Üniversitesi, Gümüşhane, Kelkit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No